CLINICAL TRIAL: NCT02671305
Title: Delivery Room Assistance With the Placental Circulation Intact: Effects on Early Postnatal Adaptation and Outcome of Preterm Babies. Study Protocol for a Randomized Control Trial (the PCI-trial)
Brief Title: Delivery Room Assistance With the Placental Circulation Intact
Acronym: PCI-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Simone Pratesi, MD, PhD, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 152-2014
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Placental Transfusion
Keywords: delayed cord clamping; cord milking; bedside neonatal resuscitation
MeSH Terms: conditions — Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placental circulation intact (Experimental): preterm newborns assisted bedside with placental circulation intact
  Interventions: Procedure: placental circulation intact
- cord milking (Active Comparator): preterm newborns who receive cord milking before assistance performed in a routine setting
  Interventions: Procedure: cord milking

INTERVENTIONS:
Procedure: placental circulation intact — bedside assistance with placental circulation intact during first 3 minutes of life
  Arms: placental circulation intact
Procedure: cord milking — neonatal assistance in a standard setting after cord milking (milking four times 20 cm of cord)
  Arms: cord milking

SUMMARY:
Preterm newborns receiving placental transfusion at birth (a volume of blood coming from the placenta towards the newborn till the cord is left unclamped) have better neonatal outcomes (in particular reduction of intraventricular hemorrhage all grade). The placental transfusion strategies performed in preterm babies at delivery have been delayed cord clamping and cord milking. Both experimental strategies do not explore the contribution of the start of breathing on placental transfusion, as performed in a small time frame (30-60 seconds for delayed clamping and less than 20 sec for cord milking). To assist the newborn bedside near to the delivering mother, leaving the cord unclamped, would allow to explore the contribution of breathing,both spontaneously started or assisted by initial steps in stabilization, on early postnatal adaptation.

The purpose of the present study is to assess the feasibility and effectiveness of delivery room assistance with the placental circulation intact in comparison to cord milking for improving outcomes in very preterm newborns.

DETAILED DESCRIPTION:
At delivery, if the cord is not clamped immediately, a volume of blood coming from the placenta continues to pass into the newborn: this placental transfusion ranges between 25 and 40 ml/kg body weight, depending on gestational age, timing of cord clamping, position of the infant at birth, onset of respirations, and administration of uterotonics to the mother. Recent research studies on animals have indicated a possible physiological role of placental transfusion in the first minutes of life, during the postnatal transition phase. During fetal life, oxygenated blood coming from the placenta through the umbilical vein largely reach the heart left ventricle through the foramen ovale. So, before birth, the placenta guarantees the left ventricle pre-load, thus maintaining cardiac output towards the aorta and epi-aortic vessels. At birth, if the cord is clamped immediately, left ventricle suddenly loose the source of its filling and the left ventricle preload becomes fully dependent on pulmonary veins return from the lungs. Pulmonary blood flow increases slowly after birth as the newly born starts breathing, in fact ventilation triggers the fall of pulmonary vascular resistances. The period between cord clamping and the onset of breathing has been indicated as "non respiring interval", when the newly born is no more receiving oxygenated blood from the placenta and not yet from the lungs. During this period, cardiac output is decreased, and hemodynamic fluctuations associated to reduced cerebral oxygenation have been demonstrated in animals. Otherwise, if the cord is maintained unclamped, blood coming from the placenta through the umbilical vein continues to fill left ventricle, while the onset of newborn's ventilation increases pulmonary blood flow and venous return. Thus, delaying cord clamping till after the start of breathing would maintain left ventricle pre-load unchanged, as demonstrated by the absence of hemodynamic fluctuations associated to reduced cerebral oxygenation in animal studies. These phenomena are probably responsible for the reduced incidence of intra-ventricular hemorrhage in babies receiving placental transfusion. Recent meta-analysis in preterm newborns demonstrated that delayed cord clamping is associated to improvement in cardiovascular stability and reduced need for inotropes, lower incidence of all grade intra-ventricular hemorrhage and necrotizing enterocolitis, lower oxygen requirement at 36 week of post-menstrual age, and less need for red blood cell transfusions, apparently without any severe short-term related morbidities or adverse effects; however, randomized trials have not yet investigated newly born infants requiring resuscitation. Placental transfusion in preterm babies may take longer, and may be incomplete if the cord is clamped within 30 to 90 seconds. This seems logical, as at term, two-thirds of the feto-placental circulation is in the infant, whilst below 30 weeks gestation, a greater proportion is in the placenta. Also, the umbilical vein is smaller than at term, and uterine contraction less efficient. Therefore, preterm babies who start breathing during a prolonged placental transfusion would probably receive the best benefits in terms of improved outcomes.

Cord milking (pinching the cord close to the mother and running the fingers towards the baby, usually 3 to 5 times) has been suggested for preterm births as a means to obtain a placental transfusion more rapidly. This procedure takes less than 20 seconds to be performed thus allowing a timely resuscitation of the newborn, in a standard setting, if needed. Cord milking over-rides the infant's physiological control of its own blood volume and blood pressure, however, and disrupts umbilical blood flow. Cord milking compared to immediate cord clamping has been recently associated in a systematic review and meta-analysis with some benefits (less oxygen requirement at 36w of gestation, and less IVH all grades) and no adverse effects in the immediate postnatal period in preterm infants less than 33 weeks of gestational age; however, further studies are warranted to assess the effect of cord milking on neonatal and long-term outcomes.

The hypothesis of the study is that to assist a preterm baby less than 30 weeks gestation with placental circulation intact allows a better postnatal adaptation and improves outcome in the neonatal period. For an ethical reason the control group will receive cord milking instead of immediate cord clamping, based on recently published results favoring cord milking in preterm babies.

The study has been designed as a two-phases study: phase 1 to assess the feasibility of the protocol (first 20 patients recruited) and phase 2 to compare the efficacy of delivery room assistance with placental circulation intact (with cord clamping at 3 minutes of life) versus cord milking for improving outcome in the neonatal period. To maximise efficiency of the planned full trial, phase 1 data would remain blind by allocated group and so would contribute to the sample size of the full trial. Recruitment of phase 1 was started on April 2016 and was completed on April 2017. Phase 1 of the study have reached the targets for feasibility. Recruitment of phase 2 (remaining 182 patients) is expected to be completed by the end of December 2018.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns with gestational age between 23+0 and 29+6 weeks
* Informed consent available

Exclusion Criteria:

* Major congenital malformation
* Hydrops fetalis, placental abruption
* Rh isoimmunization
* Twin pregnancy
* Absence of informed consent

Ages: 23 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2016-04-09 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
reduction of incidence of severe intraventricular hemorrhage, chronic lung disease or mortality | up to 36 weeks of postconceptional age
  The Outcome Measure is a composite of 3 main adverse events (severe intraventricular hemorrhage, chronic lung disease or mortality), that each patient may present or not present during the time frame. It is expected a reduction of the number of participants presenting with one or more of them. Severe intraventricular hemorrhage will be assessed by cerebral echography using Papile classification, chronic lung disease will be assessed using Jobe et al diagnostic criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Pratesi, MD, Principal Investigator — Careggi Hospital; Carlo Dani, MD, Study Director — Careggi Hospital
Locations (8):
- Italy (8):
  - UTIN-Neonatologia, Ospedale di Venere, Bari
  - UOC di Neonatologia e TIN, Dipartimento Materno-Infantile, Ospedale Maggiore, Bologna
  - Neonatal Intensive Care Unit, Department of Maternal and Infant Health, Careggi University Hospital, Florence
  - Neonatal Intensive Care Unit, IRCCS Cà Granda Foundation, Maggiore Policlinico Hospital, Milan
  - San Gerardo Hospital, Monza
  - SC TIN-Neonatologia, Azienda Ospedaliera di Perugia, Perugia
  - SOD di Neonatologia dell'Ospedale Infermi di Rimini, Rimini
  - UOC di Neonatologia e TIN, Azienda ULSS8 Berica, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pratesi S, Ciarcia M, Boni L, Ghirardello S, Germini C, Troiani S, Tulli E, Natile M, Ancora G, Barone G, Vedovato S, Bertuola F, Parata F, Mescoli G, Sandri F, Corbetta R, Ventura L, Dognini G, Petrillo F, Valenzano L, Manzari R, Lavizzari A, Mosca F, Corsini I, Poggi C, Dani C; PCI Trial Collaborators. Resuscitation With Placental Circulation Intact Compared With Cord Milking: A Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2450476. doi: 10.1001/jamanetworkopen.2024.50476. PMID 39671198
- [Derived] Pratesi S, Montano S, Ghirardello S, Mosca F, Boni L, Tofani L, Dani C. Placental Circulation Intact Trial (PCI-T)-Resuscitation With the Placental Circulation Intact vs. Cord Milking for Very Preterm Infants: A Feasibility Study. Front Pediatr. 2018 Nov 27;6:364. doi: 10.3389/fped.2018.00364. eCollection 2018. PMID 30538975